CLINICAL TRIAL: NCT02843425
Title: The Beans to Enrich the Gut Microbiome vs. Obesity's Negative Effects (BE GONE) Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0365; NCI-2016-01191 (Other: NCI CTRP)
Record Dates: First submitted 2016-07-18; First posted 2016-07-25 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer Prevention
Keywords: Cancer Prevention; Precancerous colorectal polyps; Canned beans; Questionnaires; Surveys; Stool samples
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Diet + Beans, Then Regular Diet - Beans (Experimental)
  Interventions: Other: Regular Diet; Other: Navy Beans (Canned)
- Regular Diet - Beans, Then Regular Diet + Beans (Active Comparator)
  Interventions: Other: Regular Diet; Other: Navy Beans (Canned)

INTERVENTIONS:
Other: Regular Diet — Participants follow their normal diet (not including beans for 8 weeks)
Other: Navy Beans (Canned) — Participants add 1/2 cup of canned beans per day to their diets for the first 2 weeks. This is increased to 1 cup per day for the following 6 weeks of the study.
  Other Names: Canned Beans

SUMMARY:
You are being asked to take part in this study because either you are a survivor who has a previous history of colorectal cancer or an MD Anderson patient who had a precancerous colorectal polyp or you have a previous history of colorectal cancer, and you have a current adult body mass index (BMI) score of 25 or higher.

The BMI score is used as an indicator of the level of body fat, based on height and weight.

The goal of this clinical research study is to learn if eating canned, pre-cooked beans can help improve the levels of healthy bacteria in the digestive system and reduce the effects of obesity on cancer risk.

This is an investigational study.

Up to 80 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups (intervention or control). This is done because no one knows if one study group is better, the same, or worse than the other group. Both groups will be given a diet to follow for 8 weeks.

Intervention group participants will add canned beans into their diets beginning at ½ cup per day. This will be increased to 1 cup per day during the first 2 weeks, and then will continue at 1 cup per day for the following 6 weeks of the study. You will be asked to keep a log of your bean consumption during this time.

Control group participants will be instructed to follow their normal diet (not including beans) for 8 weeks.

Length of Study:

Your active participation on the study will last a total of 20 weeks. Your participation on the study will be over after the follow-up period.

Long-Term Follow-Up:

Up to 2 times each year for up to 5 years, a member of the study staff will contact you and ask about how you are doing. You will be contacted by phone, email, or standard mail. These calls will last 15-20 minutes each.

At 6 months and 1 year after your last visit, you will complete the same questionnaires you completed at screening.

Study Visits:

At each visit, your waist measurements and weight will be collected.

Every 4 weeks (Visits 2, 3, 4, 5, and 6), blood (about 3 tablespoons) will be drawn for routine tests. You will be asked to bring a stool sample to each visit and mail a stool sample at the end of week 1 during the intervention. You will be provided with a container and instructions to collect each stool sample. You may send your stool sample back to the study staff by mail. If you choose to send it by mail, you will be given a pre-paid envelope for this.

At Visit 4, your study group assignment will be switched, and you will be assigned to the opposite group and diet from your first assignment (meaning intervention group members will be switched to the control group as well as the other way around). You will follow this new diet for the remaining 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women 30+ years of age
2. Meet criteria for overweight or obesity via BMI or waist size
3. Underwent colonoscopy screening within the past 10 years
4. History of pathology-confirmed precancerous polyp of the colon or rectum; OR Colorectal cancer survivor who has completed treatment with adequate maintenance of bowel length (eligible: hemicolectomy or low anterior resection; ineligible: total or near total colectomy, greater than 10 cm of small bowel resection) and normalized bowel habits
5. English-speaking and reside in the greater Houston/outlying areas and/or willing to travel for study-related visits at MD Anderson
6. Ability to complete web-based dietary assessments twice per week
7. Willingness to provide stool samples and undergo venipuncture
8. Willingness to consume/avoid beans as instructed during the 16 weeks from randomization

Exclusion Criteria:

1. Antibiotic use in the past month and unable/unwilling to be deferred to a later recruitment date
2. Current smoker
3. Heavy drinker (defined as more than 14 drinks per week)
4. Currently taking exclusionary prescription medications (including cytokines, immunosuppressive agents, chemopreventive drugs, bile acid sequestrants/selective cholesterol absorption inhibitors)
5. Regularly taking anti flatulence medications, probiotics and/or fiber supplements and unable/unwilling to discontinue for the purpose of the study
6. Major dietary restrictions relevant to the intervention
7. Hereditary colorectal cancer syndromes
8. Pregnant or lactating or planning to become pregnant

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Stool 16S rRNA Gene Profiles | Baseline to week 8
  The primary outcome measures will be intra- and inter-individual changes in stool 16S rRNA gene profiles at baseline, week 4 and week 8 for each cross-over period.
Changes in Blood Markers and Metabolites | Baseline to week 8
  The primary outcome measures will be intra- and inter-individual changes in blood makers and metabolites at baseline, week 8 for each cross-over period.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Daniel-MacDougall, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Zhang X, Irajizad E, Hoffman KL, Fahrmann JF, Li F, Seo YD, Browman GJ, Dennison JB, Vykoukal J, Luna PN, Siu W, Wu R, Murage E, Ajami NJ, McQuade JL, Wargo JA, Long JP, Do KA, Lampe JW, Basen-Engquist KM, Okhuysen PC, Kopetz S, Hanash SM, Petrosino JF, Scheet P, Daniel CR. Modulating a prebiotic food source influences inflammation and immune-regulating gut microbes and metabolites: insights from the BE GONE trial. EBioMedicine. 2023 Dec;98:104873. doi: 10.1016/j.ebiom.2023.104873. Epub 2023 Nov 30. PMID 38040541
- [Result] Zhang X, Browman G, Siu W, Basen-Engquist KM, Hanash SM, Hoffman KL, Okhuysen PC, Scheet P, Petrosino JF, Kopetz S, Daniel CR. The BE GONE trial study protocol: a randomized crossover dietary intervention of dry beans targeting the gut microbiome of overweight and obese patients with a history of colorectal polyps or cancer. BMC Cancer. 2019 Dec 18;19(1):1233. doi: 10.1186/s12885-019-6400-z. PMID 31852462
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org